CLINICAL TRIAL: NCT06748534
Title: Comparison of Plus Lens Addition Versus Vision Therapy for Management of Accommodative Infacility
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Superior University (Other)
Responsible Party: Principal Investigator, Muhammad Naveed Babur, Principal Investigator, Superior University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: MSRSW/Batch-Fall22/763
Record Dates: First submitted 2024-12-14; First posted 2024-12-27 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Accommodative Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interventional group I (Experimental)
  Interventions: Diagnostic Test: Plus Lens Addition (+0.75 D)
- Interventional group II (Active Comparator)
  Interventions: Combination Product: Vision Therapy Using HART Chart

INTERVENTIONS:
Diagnostic Test: Plus Lens Addition (+0.75 D) — Participants in this group were provided with +0.75 D lenses, designed to assist in alleviating strain caused by accommodative infacility by reducing the demand on the eye's focusing mechanism.
  Arms: Interventional group I
Combination Product: Vision Therapy Using HART Chart — Intervention Details: Participants in this group underwent vision therapy sessions utilizing the HART chart, aimed at enhancing their accommodative flexibility through repetitive focusing exercises.
  Arms: Interventional group II

SUMMARY:
This Randomized Control Trials Study , conducted in Lahore, Pakistan, investigates the comparative efficacy of two approaches-plus lens addition of +0.75 diopters (D) and vision therapy using the HART chart-for managing accommodative infacility. Accommodative infacility, a condition characterized by the eye's reduced ability to adjust focus between distant and near objects, impacts both visual comfort and performance, particularly during prolonged near work.

DETAILED DESCRIPTION:
The study sample comprises 38 participants, aged 15 to 35 years, divided into two groups: one group receiving plus lens addition of +0.75 D and the other undergoing structured vision therapy with the HART chart. Findings revealed that vision therapy was significantly more effective than plus lens addition, with results showing statistical significance at P < 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Participants aged 15 to 35 years.
* Diagnosed with accommodative infacility.
* Capable of adhering to the full study duration of 6 weeks.
* Measurable accommodative dysfunction confirmed through baseline eye examinations.
* Written informed consent from participants or guardians.

Exclusion Criteria:

* Presence of other significant ocular or neurological conditions.
* Inability or unwillingness to adhere to the prescribed treatment.
* Prior treatment for accommodative infacility within the past 6 months.
* Significant uncorrected refractive errors.
* Medical contraindications for using plus lenses or vision therapy.

Ages: 15 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 38 (Actual)
Dates: Start 2024-03-01 (Actual); Primary Completion 2024-08-01 (Actual); Study Completion 2025-02-28 (Estimated)

PRIMARY OUTCOMES:
Monocular and Binocular Accommodative Facility (MAF/BAF) | 12 Months
  Improvement in accommodative facility measured using Monocular and Binocular Accommodative Facility (MAF/BAF) tests with ±2.00 D flipper lenses. Measurement is recorded in cycles per minute (cpm).
subjective measures of visual comfort | 12 Months
  Reduction in symptoms of accommodative infacility assessed using a customized performa. Measurement is based on a symptom severity score recorded pre- and post-intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- Dar Ul shifa Eye Trust Hospital & Al Rehman Hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No